CLINICAL TRIAL: NCT01720186
Title: Evaluation of a Pneumotachograph (SPI) for the Production of PET and CT Acquisitions Synchronized With Breath for the Assessment of Extension of Lung Cancer
Acronym: SPI COHERENCE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 12POUM01
Record Dates: First submitted 2012-10-12; First posted 2012-11-02 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-09

CONDITIONS: Non Small Cell Lung Cancer; Lung Nodule
Keywords: Lung Cancer; PET/CT; FDG; Respiratory synchronization
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SPI Medical device (Experimental): SPI medical device used during PET/CT 4D imaging in a synchronized mode centered on the thorax.
  Interventions: Device: PET/CT 4D imaging in a synchronized mode centered on the thorax.
- reference medical device : RPM (Active Comparator): Reference medical device (RPM) used simultaneously during PET/CT 4D imaging in a synchronized mode centered on the thorax.
  Interventions: Device: PET/CT 4D imaging in a synchronized mode centered on the thorax.

INTERVENTIONS:
Device: PET/CT 4D imaging in a synchronized mode centered on the thorax.

SUMMARY:
This is a pilot study, single-center, prospective, open-label, to assess the acceptability and performance of the experimental medical device (SPI) used during an imaging examination (PET / CT 4D imaging in synchronized mode centered on the thorax). Each patient will be its own control, since the imaging examination will be synchronized simultaneously with the two systems: tested Medical Device (SPI) and reference Medical Device(RPM).

ELIGIBILITY:
Inclusion Criteria:

1. Patient for whom there is an indication of PET/CT 18FDG imaging for thoracic oncology ; this indication is consistent with the Standard Options Recommendations or was validated during Multidisciplinary Consultation Meeting :

   * Either an extension assessment of non-small cell lung cancer;
   * Either the characterization of single pulmonary nodule; Or - the definition of the target volume in radiotherapy.
2. Patient who meets the following criteria to be eligible for an PET/CT imaging:

   * Patient able to maintain a supine position for 60 minutes
   * Patient with no bronchopulmonary infection and with no upper aero digestive tract acute infection in progress (increased risk of false positives)
3. Age ≥ 18 years
4. WHO ≤ 1
5. Well-informed written consent signed by the patient and collected before any specific procedure in the study
6. Patient member in a national insurance scheme

Exclusion Criteria:

1. Patient with a bronchial carcinoid or bronchoalveolar cancer
2. Patient with acute bronchopneumopathy
3. Not stabilized diabetic patient
4. Patient with an absolute indication against spirometry: ongoing pneumothorax or within the previous month, pleural biopsy or puncture within the previous month, hemoptysis, severe asthma, tuberculosis
5. Any usual relative indication against spirometry: ongoing bronchial infections, acute asthma, decompensation of chronic respiratory failure, respiratory pain
6. Any usual formal indication against imaging examination PET/CT (important claustrophobia)
7. Patient unable to follow study procedures
8. Pregnant women or nursing mothers can not participate in the study
9. Men and women of childbearing age must use effective contraception at study entry and throughout the study
10. Any other medical conditions making the inclusion of the patient in the study inappropriate in the opinion of the investigator
11. Patient under legal guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2013-05; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Feasibility of the PET/CT synchronized exam with SPI device ("success" or "failure" ) | 2 years
  feasibility is evaluated in a composite end point (success will be obtained in case of concomitant success of the 4 sub-criteria assessment):
  1. Tolerance / acceptability of the patient to breathe into SPI throughout the examination)
  2. Detection of breath cycle of the patient by measuring dCycleSpi (dCycleSpi = Number of synchronization signals emitted by SPI / total number of breath cycle * 100).
  3. Accuracy of detection of inspiratory peak amplitudes with SPI medical device: by measuring dtSpi (dtSpi = standard deviation of the time lag between synchronization signals and maximum inspiratory amplitude for each cycle).
  4. Production of images with a correct segmentation of BTV during PET/CT synchronized exam with SPI device"

SECONDARY OUTCOMES:
Measure of dCycleRpm (dCycleRpmi = Number of synchronization signals emitted by RPM / total number of breath cycle * 100) | 2 years
Accuracy of detection of maximum inspiratory amplitudes with RPM medical device: evaluated by measuring dtRpm | 2 years
  dtRpm = standard deviation of the time lag between synchronization signals and maximum inspiratory amplitude for each cycle
Measure of BTVrpm (= biologic tumoral volume) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Frederic COURBON, PhD, Principal Investigator — Institut Claudius Regaud
Locations (1):
- Institut Claudius REGAUD, Toulouse, France